CLINICAL TRIAL: NCT00226499
Title: Study in Healthy Children (<2 Years) to Evaluate the Safety and Efficacy of GSK Biologicals' Live Attenuated Varicella Vaccine (VarilrixTM) and of GSK Biologicals' Combined Measles-Mumps-Rubella-Varicella Vaccine
Brief Title: Evaluate Vaccine Against Chickenpox and a Combined Vaccine Against 4 Viral Childhood Diseases: Measles, Mumps, Rubella and Chickenpox
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 100388; 104105 (EXT FU Y2) (Other: GSK); 103494 (EXT FU Y1) (Other: GSK); 104106 (EXT FU Y4-Y6-Y8-Y10) (Other: GSK); 2004-002676-41 (EudraCT Number)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Varicella; Chickenpox Vaccines
MeSH Terms: conditions — Chickenpox | interventions — Priorix-Tetra vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MMRV Group (Experimental): Subjects in this group received 2 doses of Priorix-Tetra vaccine, administered subcutaneously in the deltoid region of the left arm, one at Day 0 (Visit 1) and the other at Day 42 (Visit 2).
  Interventions: Biological: Priorix-tetra™
- OKAH Group (Experimental): Subjects in this group received 1 dose of Priorix at Day 0 (Visit 1) and 1 dose of Varilrix at Day 42 (Visit 2). Both vaccines were administered subcutaneously in the deltoid region of the left arm.
  Interventions: Biological: Priorix™; Biological: Varilrix™
- MMR Group (Active Comparator): Subjects in this group received 2 doses of Priorix, administered subcutaneously in the deltoid region of the left arm, one at Day 0 (Visit 1) and the other at Day 42 (Visit 2).
  Interventions: Biological: Priorix™

INTERVENTIONS:
Biological: Priorix-tetra™ — 2 doses administered subcutaneously, one at Day 0 and the other at Day 42 to subjects in MMRV Group
  Arms: MMRV Group
Biological: Priorix™ — 2 doses administered subcutaneously, one at Day 0 and the other at Day 42 to subjects in MMR Group and one dose administered subcutaneously at Day 0 to subjects in OKAH Group
  Arms: MMR Group; OKAH Group
Biological: Varilrix™ — 1 dose administered subcutaneously at Day 42 to subjects in OKAH Group
  Arms: OKAH Group

SUMMARY:
An observer-blind study to evaluate GlaxoSmithKline Biologicals' live attenuated varicella vaccine and GlaxoSmithKline Biologicals' combined measles-mumps-rubella-varicella vaccine in the prevention of varicella disease in children. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
According to treatment group allocation, participants will receive study vaccines and be followed for antibody titres and occurrence of varicella disease.

This study is conducted in 2 phases. Phase A includes the vaccination period and an observation period for efficacy. The efficacy endpoints will be evaluated over at least two years after vaccination. During this period, the immunogenicity endpoints will be evaluated with respect to the immune response 43 days after vaccination and the persistence of antibodies over two years to varicella (for all subjects) and to measles, mumps and rubella (for a subset of subjects). Regarding the safety endpoints, SAEs (including any complicated varicella cases if observed) will be assessed for all subjects during the whole Phase A duration, whereas, solicited (local and general) and unsolicited adverse events will be assessed in a subset of subjects within a 43-day period after vaccination.

Phase B is an extension of Phase A. It is a long-term follow-up until Year 10 to examine the long-term efficacy of the study vaccines against clinical varicella disease as well as the long-term persistence of antibodies to varicella (for all subjects) and to measles, mumps and rubella (in a subset of subjects) after vaccination.

ELIGIBILITY:
Inclusion criteria:

* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol for the whole duration of the study.
* Male or female subject between 12 and 22 months of age at the time of the first vaccination.
* Subjects free of obvious health problems, as established by medical history and physical examination before entering the study.
* Written informed consent obtained from the parents/guardians of the subject after they have been informed on the risks and benefits of the study, in a language they clearly understand and before performance of any study procedure.
* Subjects whose parents/guardians have direct access to telephone/mobile phone.
* Subjects:

  1. with at least one sibling (with negative history of varicella disease/vaccination) at home, or
  2. attending day care center, or
  3. attending childminders, i.e. someone taking care of several children, or
  4. who are in contact for at least once a week with other children without a known positive history of varicella disease/vaccination, while playing in close physical contact for more than 5 minutes.

Exclusion criteria:

* Previous vaccination against measles, mumps, rubella and/or varicella.
* History of previous measles, mumps, rubella and/or varicella/ herpes zoster diseases.
* Known exposure to measles, mumps, rubella and/or varicella/herpes zoster within 30 days prior to the start of the study.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of immunoglobulins and/or any blood products within three months prior to the first vaccine dose or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical.
* Family history of congenital or hereditary immunodeficiency.
* History of allergic diseases or reactions likely to be exacerbated by any component of the vaccines, including systemic allergy to egg proteins or neomycin.
* Major congenital defects or serious chronic illness.
* Residence in the same household as newborns (0-4 weeks of age), pregnant women who are varicella-susceptible, persons with a known immunodeficiency or any other persons at high risk for varicella.
* History of any neurologic disorders or seizures.
* Use of any investigational or non-registered product (drug/vaccine other than the study vaccines) within 14 days prior to vaccination and planned use during the study period.

Additional exclusion criteria for subjects included in the subset:

- Administration of a licensed vaccine within 14 days prior to vaccination and planned use until approximately 42 days after the last study vaccine dose (Day 84) with the exception of oral polio vaccine (OPV).

Ages: 11 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5803 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2006-10-12 (Actual); Study Completion 2006-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (89):
- Czechia (16):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Chomutov
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Havlíčkův Brod
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Humpolec
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kolín
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Moravská Ostrava
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Znojmo
- Greece (9):
  - GSK Investigational Site, Arta
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Giannitsá
  - GSK Investigational Site, Karditsa
  - GSK Investigational Site, Komotini
  - GSK Investigational Site, Ptolemaida
  - GSK Investigational Site, Thessaloniki
  - GSK Investigational Site, Tripoli
  - GSK Investigational Site, Véria
- Italy (9):
  - GSK Investigational Site, Quarto (NA), Campania
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Alghero (SS), Sardinia
  - GSK Investigational Site, Ozieri (SS), Sardinia
  - GSK Investigational Site, Florence, Tuscany
- Lithuania (6):
  - GSK Investigational Site, Alytus
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Panevezys
  - GSK Investigational Site, Šiauliai
  - GSK Investigational Site, Vilnius
- Norway (5):
  - GSK Investigational Site, Bekkestua
  - GSK Investigational Site, Moelv
  - GSK Investigational Site, Paradis
  - GSK Investigational Site, Skien
  - GSK Investigational Site, Trondheim
- Poland (10):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Oleśnica
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Wesoła
  - GSK Investigational Site, Wroclaw
- Romania (6):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Sibiu
  - GSK Investigational Site, Timișoara
- Russia (11):
  - GSK Investigational Site, Ivanteevka Moscow Region
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, Novokuznetsk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Volgograd
  - GSK Investigational Site, Yekaterinburg
- Slovakia (12):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Dlhá nad Oravou
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Dubnica nad Váhom
  - GSK Investigational Site, Nová Dubnica
  - GSK Investigational Site, Nové Mesto nad Váhom
  - GSK Investigational Site, Nové Zámky
  - GSK Investigational Site, Púchov
  - GSK Investigational Site, Ružomberok
  - GSK Investigational Site, Štúrovo
  - GSK Investigational Site, Šurany
  - GSK Investigational Site, Trenčín
- Sweden (5):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Norrköping
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Henry O, Brzostek J, Czajka H, Leviniene G, Reshetko O, Gasparini R, Pazdiora P, Plesca D, Desole MG, Kevalas R, Gabutti G, Povey M, Innis B. One or two doses of live varicella virus-containing vaccines: Efficacy, persistence of immune responses, and safety six years after administration in healthy children during their second year of life. Vaccine. 2018 Jan 8;36(3):381-387. doi: 10.1016/j.vaccine.2017.11.081. Epub 2017 Dec 7. PMID 29224964
- [Background] Prymula R, Bergsaker MR, Esposito S, Gothefors L, Man S, Snegova N, Stefkovicova M, Usonis V, Wysocki J, Douha M, Vassilev V, Nicholson O, Innis BL, Willems P. Protection against varicella with two doses of combined measles-mumps-rubella-varicella vaccine versus one dose of monovalent varicella vaccine: a multicentre, observer-blind, randomised, controlled trial. Lancet. 2014 Apr 12;383(9925):1313-1324. doi: 10.1016/S0140-6736(12)61461-5. Epub 2014 Jan 29. PMID 24485548
- [Background] Carryn S, Feyssaguet M, Povey M, Di Paolo E. Long-term immunogenicity of measles, mumps and rubella-containing vaccines in healthy young children: A 10-year follow-up. Vaccine. 2019 Aug 23;37(36):5323-5331. doi: 10.1016/j.vaccine.2019.07.049. Epub 2019 Jul 22. PMID 31345639
- [Derived] Habib MA, Prymula R, Carryn S, Esposito S, Henry O, Ravault S, Usonis V, Wysocki J, Gillard P, Povey M. Correlation of protection against varicella in a randomized Phase III varicella-containing vaccine efficacy trial in healthy infants. Vaccine. 2021 Jun 8;39(25):3445-3454. doi: 10.1016/j.vaccine.2021.02.074. Epub 2021 Mar 16. PMID 33736915
- [Derived] Povey M, Henry O, Riise Bergsaker MA, Chlibek R, Esposito S, Flodmark CE, Gothefors L, Man S, Silfverdal SA, Stefkovicova M, Usonis V, Wysocki J, Gillard P, Prymula R. Protection against varicella with two doses of combined measles-mumps-rubella-varicella vaccine or one dose of monovalent varicella vaccine: 10-year follow-up of a phase 3 multicentre, observer-blind, randomised, controlled trial. Lancet Infect Dis. 2019 Mar;19(3):287-297. doi: 10.1016/S1473-3099(18)30716-3. Epub 2019 Feb 11. PMID 30765242
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 100388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MMRV Group | OKAH Group | MMR Group
Started | 2489 | 2487 | 827
Completed | 1415 | 1415 | 468
Not Completed | 1074 | 1072 | 359
Not completed — Adverse Event | 10 | 6 | 3
Not completed — Others | 1064 | 1066 | 356

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMRV Group | OKAH Group | MMR Group | Total
Number analyzed (Participants) | 2489 | 2487 | 827 | 5803
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.3 (2.5) | 14.2 (2.5) | 14.2 (2.5) | 14.2 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1154 | 1223 | 401 | 2778
  Male | 1335 | 1264 | 426 | 3025
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American hispanic | 1 | 5 | 2 | 8
  Race: Arabic/north african | 24 | 7 | 3 | 34
  Race: Black | 9 | 9 | 1 | 19
  Race: East/south east asian | 8 | 7 | 1 | 16
  Race: Japanese | 1 | 0 | 0 | 1
  Race: Other | 13 | 11 | 1 | 25
  Race: South asian | 3 | 2 | 1 | 6
  Race: White/caucasian | 2430 | 2446 | 818 | 5694

OUTCOME MEASURES:

1. Primary Outcome: Phase A: Number of Subjects With Confirmed Varicella Case
Description: Confirmed varicella case = A case that met the clinical case definition [an illness with acute onset of diffuse, generalized maculopapulovesicular rash (i.e. spots, papules and/or vesicles) without other apparent cause] at least in the opinion of the investigator and was confirmed by laboratory test [Polymerase Chain Reaction (PCR) (+)] OR a case that met the clinical definition confirmed by the Independent Data Monitoring Committee (IDMC) and was epidemiologically linked [Epi (+)] to a valid index case.
Time Frame: From 42 days post dose 2 until the end of Phase A
Population: The analysis was performed on the According-to-Protocol (ATP) Cohort for Efficacy (Phase A), which included all evaluable subjects who had efficacy follow-up starting from 42 days post dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 2279 | 2263 | 743
Participants | 37 | 243 | 201
Statistical Analysis 1: Comparison: MMRV Group vs MMR Group; Vaccine Efficacy (VE) was measured by calculating the relative risk of a confirmed varicella case in a vaccine group compared to a confirmed varicella case in the control group; Test type: Other — To demonstrate at least 60% VE, with respect to confirmed varicella disease over at least a two-year period of follow-up (beginning 42 days post dose 2) of Priorix-Tetra as compared to Priorix); p < 0.0001, Regression, Cox; Vaccine Efficacy = 94.943, 97.5% CI 2-sided [92.446 to 96.615]
Statistical Analysis 2: Comparison: OKAH Group vs MMR Group; [analysis description as in outcome 1, analysis 1]; Test type: Other — To demonstrate at least 60% VE, with respect to confirmed varicella disease over at least a two-year period of follow-up (beginning 42 days post dose 2) of Varilrix as compared to Priorix); p = 0.1265, Regression, Cox; Vaccine Efficacy = 65.428, 97.5% CI 2-sided [57.182 to 72.086]

2. Secondary Outcome: Phase A: Number of Subjects With Moderate or Severe Confirmed Varicella Case
Description: Confirmed varicella case: A case that met the clinical case definition at least in the opinion of the investigator and was confirmed by laboratory test [PCR (+)] OR a case that met the clinical definition confirmed by the IDMC and was epidemiologically linked [Epi (+)] to a valid index case. Moderately severe disease: 8-15 points; severe disease: ≥ 16 points (scored by IDMC using the modified Vázquez scale).
Time Frame: From 42 days post dose 2 until the end of Phase A
Population: The analysis was performed on the ATP Cohort for Efficacy (Phase A), which included all evaluable subjects who had efficacy follow-up starting from 42 days post dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 2279 | 2263 | 743
Participants | 2 | 37 | 117
Statistical Analysis 1: Comparison: MMRV Group vs MMR Group; VE was measured by calculating the relative risk of a moderate or severe confirmed varicella case in a vaccine group compared to a moderate or severe confirmed varicella case in the control group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0001, Regression, Cox; Vaccine Efficacy = 99.498, 95% CI 2-sided [97.522 to 99.898]
Statistical Analysis 2: Comparison: OKAH Group vs MMR Group; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.1265, Regression, Cox; Vaccine Efficacy = 90.741, 95% CI 2-sided [85.866 to 93.934]

3. Secondary Outcome: Phase A: Number of Subjects With Probable or Confirmed Varicella Case
Description: Probable or confirmed varicella case = A case that met the clinical case definition (as determined by the IDMC) but was not laboratory confirmed [PCR (-)] AND was not epidemiologically linked [Epi (-)] to another probable or confirmed case.
Time Frame: From 42 days post dose 2 until the end of Phase A
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 2279 | 2263 | 743
Participants | 57 | 260 | 209
Statistical Analysis 1: Comparison: MMRV Group vs MMR Group; VE was measured by calculating the relative risk of a probable or confirmed varicella case in a vaccine group compared to a probable or confirmed varicella case in the control group; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Cox; Vaccine Efficacy = 92.487, 95% CI 2-sided [89.927 to 94.396]
Statistical Analysis 2: Comparison: OKAH Group vs MMR Group; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.1265, Regression, Cox; Vaccine Efficacy = 64.585, 95% CI 2-sided [57.503 to 70.486]

4. Secondary Outcome: Phase A: Immune Response to Varicella Vaccine With Respect to Anti-Varicella Zoster Virus (Anti-VZV) Antibody Concentrations
Description: Anti-VZV antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in milliinternational units per milliliter (mIU/mL).
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: The analysis was performed on the ATP Cohort for Immunogenicity, which included all evaluable subjects who had pre-vaccination results available for at least one of the vaccine components.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 2245 | 2245 | 742
mIU/mL
  Anti-VZV, Day 0 | 12.8 [12.6 to 12.9] | 12.7 [12.6 to 12.8] | 12.6 [12.5 to 12.8]
  Anti-VZV, Day 42: number analyzed (Participants) | 690 | 697 | 231
  Anti-VZV, Day 42 | 116.1 [108.3 to 124.5] | 13.5 [13.0 to 14.1] | 13.1 [12.5 to 13.9]
  Anti-VZV, Day 84: number analyzed (Participants) | 2241 | 2234 | 740
  Anti-VZV, Day 84 | 1833.3 [1767.8 to 1901.3] | 98.1 [94.2 to 102.3] | 14.7 [13.9 to 15.6]
  Anti-VZV, Year 1: number analyzed (Participants) | 2066 | 2053 | 673
  Anti-VZV, Year 1 | 365.1 [349.0 to 381.9] | 145.2 [137.0 to 153.8] | 20.3 [18.2 to 22.5]
  Anti-VZV, Year 2: number analyzed (Participants) | 1924 | 1916 | 635
  Anti-VZV, Year 2 | 414.6 [392.1 to 438.5] | 170.6 [158.1 to 184.1] | 36.9 [31.6 to 43.1]

5. Secondary Outcome: Phase A: Number of Subjects With Seroconversion/Seroresponse to VZV
Description: Seronegative (S-) = Subjects with antibody concentration less than (<) 25 mIU/mL prior to vaccination. Seropositive (S+) = Subjects with antibody concentration greater than or equal to (≥) 25 mIU/mL prior to vaccination. Seroconversion was defined as the appearance of antibodies (i.e. titer greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination.
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 2245 | 2245 | 742
Participants
  Anti-VZV, Day 0 | 26 | 24 | 4
  Anti-VZV, Day 42: number analyzed (Participants) | 690 | 697 | 231
  Anti-VZV, Day 42 | 661 | 21 | 6
  Anti-VZV, Day 84: number analyzed (Participants) | 2241 | 2234 | 740
  Anti-VZV, Day 84 | 2236 | 2123 | 40
  Anti-VZV, Year 1: number analyzed (Participants) | 2066 | 2053 | 673
  Anti-VZV, Year 1 | 2056 | 1968 | 91
  Anti-VZV, Year 2: number analyzed (Participants) | 1924 | 1916 | 635
  Anti-VZV, Year 2 | 1913 | 1776 | 170

6. Secondary Outcome: Phase A: Immune Response to Measles With Respect to Anti-measles Antibody Concentrations in a Subset of Subjects
Description: Anti-measles antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in milliinternational units per milliliter (mIU/mL).
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 704 | 713 | 232
mIU/mL
  Anti-measles, Day 0 | 75.7 [74.6 to 76.8] | 77.9 [75.6 to 80.3] | 77.9 [73.9 to 82.1]
  Anti-measles, Day 42: number analyzed (Participants) | 691 | 698 | 230
  Anti-measles, Day 42 | 3961.0 [3719.7 to 4217.9] | 2602.7 [2429.6 to 2788.1] | 2817.4 [2506.3 to 3167.1]
  Anti-measles, Day 84: number analyzed (Participants) | 704 | 712 | 231
  Anti-measles, Day 84 | 5809.6 [5544.5 to 6087.3] | 3438.1 [3210.9 to 3681.5] | 3695.0 [3318.2 to 4114.6]
  Anti-measles, Year 1: number analyzed (Participants) | 630 | 630 | 200
  Anti-measles, Year 1 | 4993.7 [4714.7 to 5289.2] | 2856.8 [2658.6 to 3069.7] | 2885.7 [2520.7 to 3303.5]
  Anti-measles, Year 2: number analyzed (Participants) | 589 | 593 | 187
  Anti-measles, Year 2 | 4709.6 [4407.1 to 5033.0] | 2624.5 [2423.6 to 2842.2] | 2677.9 [2302.5 to 3114.5]

7. Secondary Outcome: Phase A: Number of Subjects With Seroconversion/Seroresponse to Measles in a Subset of Subjects
Description: Seronegative (S-) = Subjects with antibody concentration < 150 mIU/mL prior to vaccination. Seropositive (S+) = Subjects with antibody concentration ≥ 150 mIU/mL prior to vaccination. Seroconversion was defined as the appearance of antibodies (i.e. titer greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination.
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 704 | 713 | 232
Participants
  Anti-measles, Day 0 | 2 | 7 | 2
  Anti-measles, Day 42: number analyzed (Participants) | 691 | 698 | 230
  Anti-measles, Day 42 | 676 | 682 | 225
  Anti-measles, Day 84: number analyzed (Participants) | 704 | 712 | 231
  Anti-measles, Day 84 | 703 | 702 | 230
  Anti-measles, Year 1: number analyzed (Participants) | 630 | 630 | 200
  Anti-measles, Year 1 | 628 | 621 | 198
  Anti-measles, Year 2: number analyzed (Participants) | 589 | 593 | 187
  Anti-measles, Year 2 | 584 | 583 | 183

8. Secondary Outcome: Phase A: Immune Response to Mumps With Respect to Anti-mumps Antibody Concentrations in a Subset of Subjects
Description: Anti-mumps antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in units per milliliter (U/mL).
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 704 | 712 | 232
U/mL
  Anti-mumps, Day 0 | 117.5 [115.4 to 119.7] | 119.1 [116.2 to 122.2] | 118.1 [114.4 to 122.0]
  Anti-mumps, Day 42: number analyzed (Participants) | 667 | 670 | 225
  Anti-mumps, Day 42 | 896.6 [827.0 to 972.0] | 925.0 [859.4 to 995.7] | 945.2 [839.0 to 1064.9]
  Anti-mumps, Day 84: number analyzed (Participants) | 698 | 701 | 225
  Anti-mumps, Day 84 | 1496.8 [1407.7 to 1591.7] | 759.8 [705.5 to 818.3] | 1547.9 [1408.0 to 1701.6]
  Anti-mumps, Year 1: number analyzed (Participants) | 624 | 622 | 196
  Anti-mumps, Year 1 | 1008.6 [928.8 to 1095.2] | 875.9 [805.8 to 952.2] | 1089.6 [944.0 to 1257.5]
  Anti-mumps, Year 2: number analyzed (Participants) | 582 | 587 | 187
  Anti-mumps, Year 2 | 1050.6 [957.5 to 1152.7] | 882.0 [805.6 to 965.6] | 989.4 [848.3 to 1153.9]

9. Secondary Outcome: Phase A: Number of Subjects With Seroconversion/Seroresponse to Mumps in a Subset of Subjects
Description: Seronegative (S-) = Subjects with antibody concentration < 231 U/mL prior to vaccination. Seropositive (S+) = Subjects with antibody concentration ≥ 231 U/mL prior to vaccination. Seroconversion was defined as the appearance of antibodies (i.e. titer greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination.
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 704 | 712 | 232
Participants
  Anti-mumps, Day 0 | 4 | 6 | 2
  Anti-mumps, Day 42: number analyzed (Participants) | 667 | 670 | 225
  Anti-mumps, Day 42 | 584 | 613 | 208
  Anti-mumps, Day 84: number analyzed (Participants) | 698 | 701 | 225
  Anti-mumps, Day 84 | 683 | 608 | 225
  Anti-mumps, Year 1: number analyzed (Participants) | 624 | 622 | 196
  Anti-mumps, Year 1 | 569 | 554 | 182
  Anti-mumps, Year 2: number analyzed (Participants) | 582 | 587 | 187
  Anti-mumps, Year 2 | 527 | 520 | 171

10. Secondary Outcome: Phase A: Immune Response to Rubella With Respect to Anti-rubella Antibody Concentrations in a Subset of Subjects
Description: Anti-rubella antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in International Units per milliliter (IU/mL).
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 704 | 713 | 232
IU/mL
  Anti-rubella, Day 0 | 2.1 [2.0 to 2.1] | 2.0 [2.0 to 2.1] | 2.1 [2.0 to 2.2]
  Anti-rubella, Day 42: number analyzed (Participants) | 692 | 698 | 230
  Anti-rubella, Day 42 | 57.6 [54.2 to 61.2] | 74.0 [69.9 to 78.3] | 71.0 [64.8 to 77.8]
  Anti-rubella, Day 84: number analyzed (Participants) | 704 | 712 | 231
  Anti-rubella, Day 84 | 104.7 [99.8 to 109.8] | 122.1 [116.2 to 128.2] | 111.9 [103.5 to 120.9]
  Anti-rubella, Year 1: number analyzed (Participants) | 630 | 630 | 200
  Anti-rubella, Year 1 | 88.7 [83.9 to 93.8] | 103.7 [97.8 to 110.0] | 98.0 [88.7 to 108.3]
  Anti-rubella, Year 2: number analyzed (Participants) | 589 | 593 | 187
  Anti-rubella, Year 2 | 71.8 [67.5 to 76.4] | 79.1 [74.2 to 84.3] | 71.8 [64.0 to 80.5]

11. Secondary Outcome: Phase A: Number of Subjects With a Seroconversion/Seroresponse to Rubella in a Subset of Subjects
Description: Seronegative (S-) = Subjects with antibody concentration < 4 IU/mL prior to vaccination. Seropositive (S+) = Subjects with antibody concentration ≥ 4 IU/mL prior to vaccination. Seroconversion was defined as the appearance of antibodies (i.e. titer greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination.
Time Frame: At Day 0, Day 42, Day 84, Year 1 and Year 2 time points
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 704 | 713 | 232
Participants
  Anti-rubella, Day 0 | 7 | 5 | 2
  Anti-rubella, Day 42: number analyzed (Participants) | 692 | 698 | 230
  Anti-rubella, Day 42 | 688 | 693 | 230
  Anti-rubella, Day 84: number analyzed (Participants) | 704 | 712 | 231
  Anti-rubella, Day 84 | 704 | 710 | 231
  Anti-rubella, Year 1: number analyzed (Participants) | 630 | 630 | 200
  Anti-rubella, Year 1 | 630 | 628 | 200
  Anti-rubella, Year 2: number analyzed (Participants) | 589 | 593 | 187
  Anti-rubella, Year 2 | 589 | 590 | 186

12. Secondary Outcome: Phase A: Number of Subjects With Confirmed Cases of Herpes Zoster
Description: The number of subjects with confirmed cases of herpes zoster is reported.
Time Frame: From Day 0 until the end of Phase A (Year 2)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 807 | 812 | 268
Participants | 0 | 0 | 0

13. Secondary Outcome: Phase A: Number of Subjects Reporting Fever
Description: All fever = Occurrence of any fever (measured rectally) regardless of its intensity grade or relationship to vaccination. Related = fever (measured rectally) assessed by the investigator to be causally related to the study vaccination. Medical Advice = seek for medical advice.
Time Frame: Within 43 days (Day 0-42) post-vaccination period following each dose
Population: The analysis was performed on a subset of the Total Vaccinated Cohort. The subset of subjects was identified as 200 subjects from each country. Depending on the country, this subset was stipulated to be either the first 200 subjects enrolled irrespective of the study center or 200 subjects enrolled at selected centers.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 784 | 795 | 256
Participants
  All Fever, Dose 1 | 503 | 439 | 132
  Related Fever, Dose 1 | 332 | 240 | 82
  Related Fever ≥ 38°C, Dose 1 | 332 | 240 | 82
  Related Fever > 38.5°C, Dose 1 | 222 | 147 | 46
  Related Fever > 39°C, Dose 1 | 141 | 90 | 29
  Related Fever > 39.5°C, Dose 1 | 71 | 48 | 13
  Related Fever > 40°C, Dose 1 | 22 | 18 | 5
  Fever ≥ 38°C, Dose 1 | 503 | 439 | 132
  Fever > 38.5°C, Dose 1 | 359 | 297 | 84
  Fever > 39°C, Dose 1 | 249 | 191 | 55
  Fever > 39.5°C, Dose 1 | 139 | 100 | 29
  Fever > 40°C, Dose 1 | 49 | 43 | 15
  Fever Medical Advice, Dose 1 | 203 | 177 | 46
  All Fever, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  All Fever, Dose 2 | 303 | 313 | 103
  Related Fever, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever, Dose 2 | 136 | 144 | 41
  Related Fever ≥ 38°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever ≥ 38°C, Dose 2 | 136 | 144 | 41
  Related Fever > 38.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 38.5°C, Dose 2 | 78 | 88 | 25
  Related Fever > 39°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 39°C, Dose 2 | 51 | 54 | 20
  Related Fever > 39.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 39.5°C, Dose 2 | 25 | 32 | 11
  Related Fever > 40°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 40°C, Dose 2 | 9 | 9 | 3
  Fever ≥ 38°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever ≥ 38°C, Dose 2 | 303 | 313 | 103
  Fever > 38.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 38.5°C, Dose 2 | 212 | 205 | 69
  Fever > 39°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 39°C, Dose 2 | 136 | 132 | 54
  Fever > 39.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 39.5°C, Dose 2 | 66 | 74 | 30
  Fever > 40°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 40°C, Dose 2 | 20 | 25 | 8
  Fever Medical Advice, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever Medical Advice, Dose 2 | 112 | 119 | 44

14. Secondary Outcome: Phase A: Number of Subjects Reporting Fever
Description: All fever = Occurrence of any fever (measured rectally) regardless of its intensity grade or relationship to vaccination. Related fever = fever (measured rectally) assessed by the investigator to be causally related to the study vaccination. Medical Advice = seek for medical advice.
Time Frame: Within 15 days (Day 0-14) post-vaccination period following each dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 784 | 795 | 256
Participants
  All Fever, Dose 1 | 450 | 354 | 102
  Related Fever, Dose 1 | 328 | 226 | 69
  Related Fever ≥ 38°C, Dose 1 | 328 | 226 | 69
  Related Fever > 38.5°C, Dose 1 | 216 | 134 | 36
  Related Fever > 39°C, Dose 1 | 135 | 82 | 23
  Related Fever > 39.5°C, Dose 1 | 67 | 42 | 10
  Related Fever > 40°C, Dose 1 | 19 | 15 | 4
  Fever ≥ 38°C, Dose 1 | 449 | 349 | 101
  Fever > 38.5°C, Dose 1 | 300 | 213 | 54
  Fever > 39°C, Dose 1 | 196 | 124 | 34
  Fever > 39.5°C, Dose 1 | 101 | 58 | 16
  Fever > 40°C, Dose 1 | 30 | 21 | 6
  Fever Medical Advice, Dose 1 | 140 | 100 | 26
  All Fever, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  All Fever, Dose 2 | 189 | 201 | 55
  Related Fever, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever, Dose 2 | 118 | 125 | 32
  Related Fever ≥ 38°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever ≥ 38°C, Dose 2 | 118 | 125 | 32
  Related Fever > 38.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 38.5°C, Dose 2 | 60 | 73 | 18
  Related Fever > 39°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 39°C, Dose 2 | 34 | 41 | 16
  Related Fever > 39.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 39.5°C, Dose 2 | 17 | 22 | 9
  Related Fever > 40°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Fever > 40°C, Dose 2 | 6 | 5 | 3
  Fever ≥ 38°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever ≥ 38°C, Dose 2 | 184 | 200 | 51
  Fever > 38.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 38.5°C, Dose 2 | 101 | 110 | 30
  Fever > 39°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 39°C, Dose 2 | 62 | 65 | 24
  Fever > 39.5°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 39.5°C, Dose 2 | 28 | 35 | 14
  Fever > 40°C, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever > 40°C, Dose 2 | 8 | 11 | 4
  Fever Medical Advice, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Fever Medical Advice, Dose 2 | 43 | 48 | 13

15. Secondary Outcome: Phase A: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any solicited local symptom = Occurrence of any local symptom regardless of their intensity grade. Grade 3 pain = Cried when limb was moved/spontaneously painful. Grade 3 redness and swelling = greater than (>) 20 mm.
Time Frame: 4 days post-vaccination period following each dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 782 | 796 | 256
Participants
  Any Pain, Dose 1 | 74 | 83 | 20
  Grade 3 Pain, Dose 1 | 1 | 2 | 0
  Any Redness, Dose 1 | 137 | 154 | 36
  Grade 3 Redness, Dose 1 | 3 | 3 | 0
  Any Swelling, Dose 1 | 38 | 37 | 6
  Grade 3 Swelling, Dose 1 | 3 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 758 | 774 | 247
  Any Pain, Dose 2 | 91 | 63 | 16
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 758 | 774 | 247
  Grade 3 Pain, Dose 2 | 0 | 1 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 758 | 774 | 247
  Any Redness, Dose 2 | 188 | 106 | 23
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 758 | 774 | 247
  Grade 3 Redness, Dose 2 | 26 | 3 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 758 | 774 | 247
  Any Swelling, Dose 2 | 72 | 31 | 3
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 758 | 774 | 247
  Grade 3 Swelling, Dose 2 | 4 | 0 | 0

16. Secondary Outcome: Phase A: Number of Subjects Reporting Meningism
Description: Any = Occurrence of meningism regardless of its intensity grade. Grade 3 meningism = Prevented normal, everyday activities. Related = Assessed by the investigator to be causally related to the study vaccination.
Time Frame: Within 43 days (Day 0-42) post-vaccination period following each dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 784 | 795 | 256
Participants
  Any Meningism, Dose 1 | 1 | 0 | 0
  Grade 3 Meningism, Dose 1 | 1 | 0 | 0
  Related Meningism, Dose 1 | 1 | 0 | 0
  Any Meningism, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Any Meningism, Dose 2 | 0 | 1 | 0
  Grade 3 Meningism, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Grade 3 Meningism, Dose 2 | 0 | 0 | 0
  Related Meningism, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Meningism, Dose 2 | 0 | 0 | 0

17. Secondary Outcome: Phase A: Number of Subjects Reporting Parotitis
Description: Any = Occurrence of parotitis regardless of its intensity grade. Grade 3 parotitis = Swelling with accompanying general symptoms. Related = Assessed by the investigator to be causally related to the study.
Time Frame: Within 43 days (Day 0-42) post-vaccination period following each dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 784 | 795 | 256
Participants
  Any Parotitis, Dose 1 | 4 | 5 | 1
  Grade 3 Parotitis, Dose 1 | 2 | 1 | 0
  Related Parotitis, Dose 1 | 3 | 3 | 0
  Any Parotitis, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Any Parotitis, Dose 2 | 0 | 2 | 0
  Grade 3 Parotitis, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Grade 3 Parotitis, Dose 2 | 0 | 1 | 0
  Related Parotitis, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Related Parotitis, Dose 2 | 0 | 1 | 0

18. Secondary Outcome: Phase A: Number of Subjects Reporting Rash
Description: Any = Occurrence of rash regardless of its intensity grade. Grade 3 rash = 101-500 lesions. Grade 4 rash = > 500 lesions. Related rash = Assessed by the investigator to be causally related to the study vaccination.
Time Frame: Within 43 days (Day 0-42) post-vaccination period following each dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 784 | 795 | 256
Participants
  Any Localized or Generalized,Dose 1 | 82 | 84 | 30
  Any Localized, Dose 1 | 14 | 15 | 6
  Localized Admin. site, Dose 1 | 0 | 1 | 0
  Localized Other site, Dose 1 | 14 | 14 | 6
  Any Generalized, Dose 1 | 68 | 69 | 24
  Generalized With fever, Dose 1 | 41 | 41 | 14
  Generalized Measles/Rubella, Dose 1 | 30 | 24 | 9
  Generalized Grade 3/4, Dose 1 | 9 | 12 | 7
  Generalized Grade 4, Dose 1 | 2 | 2 | 4
  Generalized Related, Dose 1 | 27 | 32 | 13
  Any Localized or Generalized,Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Any Localized or Generalized,Dose 2 | 42 | 36 | 9
  Any Localized, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Any Localized, Dose 2 | 5 | 12 | 4
  Localized Admin. site, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Localized Admin. site, Dose 2 | 0 | 2 | 0
  Localized Other site, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Localized Other site, Dose 2 | 5 | 10 | 4
  Any Generalized, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Any Generalized, Dose 2 | 37 | 24 | 5
  Generalized With fever, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Generalized With fever, Dose 2 | 9 | 11 | 4
  Generalized Measles/Rubella, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Generalized Measles/Rubella, Dose 2 | 8 | 4 | 0
  Generalized Grade 3/4, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Generalized Grade 3/4, Dose 2 | 5 | 6 | 1
  Generalized Grade 4, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Generalized Grade 4, Dose 2 | 2 | 1 | 0
  Generalized Related, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Generalized Related, Dose 2 | 12 | 6 | 1

19. Secondary Outcome: Phase A: Number of Subjects With Suspected Sign of Meningism Including Febrile Convulsions
Description: Any = Occurrence of meningism including febrile convulsions regardless of intensity grade.
Time Frame: Within 43 days (Day 0-42) post-vaccination period following each dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 784 | 795 | 256
Participants
  Meningism including febrile convulsions, Dose 1 | 1 | 0 | 0
  Meningism including febrile convulsions, Dose 2: number analyzed (Participants) | 758 | 773 | 247
  Meningism including febrile convulsions, Dose 2 | 0 | 1 | 0

20. Secondary Outcome: Phase A: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE assessed included any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = Occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: Within 43 days (Day 0-42) post-vaccination period following each dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 807 | 812 | 268
Participants
  Any AE(s), Dose 1 | 301 | 303 | 82
  Any AE(s), Dose 2: number analyzed (Participants) | 777 | 788 | 253
  Any AE(s), Dose 2 | 239 | 258 | 90

21. Secondary Outcome: Phase A: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life-threatening, required hospitalisation or prolongation of hospitalisation or resulted in disability/incapacity. Any SAE = occurrence of SAE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 until the end of Phase A (Year 2)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 2489 | 2487 | 827
Participants | 473 | 480 | 148

22. Secondary Outcome: Phase A: Health Economics Analysis of Factors Leading to Indirect Costs Due to Varicella Illness
Description: Parameters assessed: 1. Number of hours lost from work by parents/guardians as a result of taking care of their child due to varicella. 2. Number of hours the child lost attendance in: day care/childminder, school, or in any extra-curricular activities (e.g. sports or recreation or any type of organised leisure activities) due to varicella. 3. Number of hours spent by a nurse, a babysitter or any type of existing paid caregiver to look after the child (if applicable).
Time Frame: During Phase A (from Day 0 up to Year 2)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 37 | 246 | 201
Hours
  Time lost from work [hours] | 31.5 (22.9) | 40.5 (31.4) | 48.1 (35.3)
  Time lost for subjects [hours] | 66.4 (86.0) | 49.5 (31.9) | 54.5 (36.4)
  Time of requested assistance [hours] | 34.0 (31.1) | 35.2 (51.6) | 35.4 (31.3)

23. Secondary Outcome: Phase B: Number of Subjects With Confirmed Varicella Case
Description: Confirmed varicella case = A case that met the clinical case definition at least in the opinion of the investigator and was confirmed by laboratory test [PCR (+)] OR a case that met the clinical definition confirmed by the IDMC and was epidemiologically linked [Epi (+)] to a valid index case.
Time Frame: From the beginning of Phase B (Year 2) up to study end (Year 10)
Population: The analysis was performed on the ATP Cohort for Efficacy (Phase B), which included all evaluable subjects who had efficacy follow-up from the period when Phase A was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 1800 | 1591 | 396
Participants | 38 | 225 | 149
Statistical Analysis 1: Comparison: MMRV Group vs MMR Group; VE was measured by calculating the relative risk of a confirmed varicella case in a vaccine group compared to a confirmed varicella case in the control group; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Cox; Vaccine Efficacy = 95.855, 95% CI 2-sided [94.075 to 97.101]
Statistical Analysis 2: Comparison: OKAH Group vs MMR Group; [analysis description as in outcome 23, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.1265, Regression, Cox; Vaccine Efficacy = 69.812, 95% CI 2-sided [62.848 to 75.470]

24. Secondary Outcome: Phase B: Number of Subjects With Moderate or Severe Confirmed Varicella Case
Description: Confirmed varicella case = A case that met the clinical case definition at least in the opinion of the investigator and was confirmed by laboratory test [PCR (+)] OR a case that met the clinical definition confirmed by the IDMC and was epidemiologically linked [Epi (+)] to a valid index case. Moderately severe disease = 8-15 points; severe disease: ≥ 16 points (scored by IDMC using the modified Vázquez scale).
Time Frame: From the beginning of Phase B (Year 2) up to study end (Year 10)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 2279 | 2266 | 744
Participants | 6 | 67 | 176
Statistical Analysis 1: Comparison: MMRV Group vs MMR Group; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Cox; Vaccine Efficacy = 99.072, 95% CI 2-sided [97.907 to 99.589]
Statistical Analysis 2: Comparison: OKAH Group vs MMR Group; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.1265, Regression, Cox; Vaccine Efficacy = 89.532, 95% CI 2-sided [86.126 to 92.102]

25. Secondary Outcome: Phase B: Number of Subjects With Probable or Confirmed Varicella Case
Description: Probable or confirmed varicella = A case that met the clinical case definition (as determined by the IDMC) but was not laboratory confirmed [PCR (-)] AND was not epidemiologically linked [Epi (-)] to another probable or confirmed case.
Time Frame: From the beginning of Phase B (Year 2) up to study end (Year 10)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 1800 | 1591 | 396
Participants | 49 | 237 | 152
Statistical Analysis 1: Comparison: MMRV Group vs MMR Group; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Cox; Vaccine Efficacy = 94.816, 95% CI 2-sided [92.838 to 96.248]
Statistical Analysis 2: Comparison: OKAH Group vs MMR Group; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.1265, Regression, Cox; Vaccine Efficacy = 68.932, 95% CI 2-sided [61.893 to 74.671]

26. Secondary Outcome: Phase B: Characteristics of Varicella Cases
Description: Varicella cases were characterized by type, number and character of lesions, duration of rash, incidence of fever, systemic signs, the assessment by investigator, complications, treatment, outcome and intensity of severity.
Time Frame: From the beginning of Phase B (Year 2) up to study end (Year 10)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 38 | 225 | 149
Participants
  Number of varicella cases by subject, 1 | 38 | 223 | 148
  Number of varicella cases by subject, 2 | 0 | 2 | 1
  Varicella type, Any | 38 | 225 | 149
  Varicella type, Confirmed | 38 | 225 | 149
  Varicella type, Confirmed PCR | 31 | 207 | 140
  Varicella type, Confirmed EPI | 7 | 18 | 9
  Varicella type, Confirmed or Probable | 38 | 225 | 149
  Varicella type, No case | 0 | 0 | 0
  Rash: number of lesions, 1-50 | 32 | 173 | 76
  Rash: number of lesions, 51-100 | 5 | 35 | 39
  Rash: number of lesions, 101-500 | 1 | 15 | 27
  Rash: number of lesions, 501+ | 0 | 0 | 7
  Rash: number of lesions, Missing | 0 | 2 | 0
  Character of most lesions, Macular | 4 | 6 | 1
  Character of most lesions, Papular | 16 | 108 | 63
  Character of most lesions, Vesicular | 16 | 100 | 81
  Character of most lesions, Haemorragic | 2 | 6 | 4
  Character of most lesions, Missing | 0 | 5 | 0
  Duration of rash, 0 days | 0 | 0 | 0
  Duration of rash, 1-5 days | 23 | 140 | 68
  Duration of rash, 6-10 days | 10 | 67 | 61
  Duration of rash, 11-15 days | 5 | 13 | 19
  Duration of rash, 16+ days | 0 | 0 | 0
  Duration of rash, Missing | 0 | 5 | 1
  Max. number of lesions [investigator], 1-50 | 32 | 173 | 76
  Max. number of lesions [investigator], 51-100 | 5 | 35 | 39
  Max. number of lesions [investigator], 101-500 | 1 | 15 | 27
  Max. number of lesions [investigator], 501+ | 0 | 0 | 7
  Max. number of lesions [investigator], Missing | 0 | 2 | 0
  Fever, No fever | 37 | 212 | 100
  Fever, 38.8°C to 39.9°C | 1 | 13 | 43
  Fever, 40+ °C | 0 | 0 | 6
  Systemic sign, Pain in back or abdomen | 6 | 27 | 27
  Systemic sign, Interstitial pneumonia | 0 | 0 | 0
  Systemic sign, Encephalitis | 0 | 0 | 0
  Assessment by investigator, Does not appear ill | 28 | 159 | 62
  Assessment by investigator, Moderately ill | 10 | 64 | 80
  Assessment by investigator, Severely ill | 0 | 1 | 6
  Assessment by investigator, Missing | 0 | 1 | 1
  Complications, Yes | 0 | 0 | 0
  Complications, No | 38 | 222 | 147
  Complications, Missing | 0 | 3 | 2
  Treatment, Yes | 15 | 115 | 91
  Treatment, No | 23 | 106 | 56
  Treatment, Missing | 0 | 4 | 2
  Outcome, Recovered/resolved | 38 | 224 | 148
  Outcome, Recovered/resolved with sequelae | 0 | 0 | 0
  Outcome, Missing | 0 | 1 | 1
  Intensity of severity, Mild | 34 | 198 | 91
  Intensity of severity, Moderately severe | 4 | 27 | 54
  Intensity of severity, Severe | 0 | 0 | 4

27. Secondary Outcome: Phase B: Immune Response to Varicella Vaccine With Respect to Anti-Varicella Zoster Virus (Anti-VZV) Antibody Concentrations
Description: as for outcome 4
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: The analysis was performed on the Adapted persistence cohort (Adapted ATP cohort for each specific time point).
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 1342 | 1142 | 242
mIU/mL
  Anti-VZV, Year 4 | 501.3 [467.8 to 537.1] | 272.7 [246.2 to 302.1] | 32.4 [26.1 to 40.4]
  Anti-VZV, Year 6: number analyzed (Participants) | 1292 | 1021 | 176
  Anti-VZV, Year 6 | 680.6 [635.7 to 728.8] | 417.6 [379.9 to 459.0] | 91.8 [66.3 to 126.9]
  Anti-VZV, Year 8: number analyzed (Participants) | 1146 | 828 | 117
  Anti-VZV, Year 8 | 512.5 [480.3 to 546.8] | 418.5 [383.2 to 457.1] | 146.9 [99.6 to 216.6]
  Anti-VZV, Year 10: number analyzed (Participants) | 1169 | 831 | 111
  Anti-VZV, Year 10 | 471.3 [443.2 to 501.2] | 404.6 [373.0 to 438.8] | 219.6 [149.2 to 323.3]

28. Secondary Outcome: Phase B: Number of Subjects With Anti-VZV Antibody Concentrations Above the Cut-off Value
Description: The anti-VZV antibody concentration cut-off value assessed was greater than or equal to (≥) 25 mIU/mL, in the sera of subjects seronegative before vaccination.
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: The analysis was performed on the Adapted persistence cohort (Adapted ATP cohort for each specific time point).
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 1342 | 1142 | 242
Participants
  Anti-VZV, Year 4 | 1330 | 1061 | 73
  Anti-VZV, Year 6: number analyzed (Participants) | 1292 | 1021 | 176
  Anti-VZV, Year 6 | 1289 | 986 | 97
  Anti-VZV, Year 8: number analyzed (Participants) | 1146 | 828 | 117
  Anti-VZV, Year 8 | 1142 | 806 | 78
  Anti-VZV, Year 10: number analyzed (Participants) | 1169 | 831 | 111
  Anti-VZV, Year 10 | 1164 | 818 | 81

29. Secondary Outcome: Phase B: Immune Response to Measles With Respect to Anti-measles Antibody Concentrations
Description: as for outcome 6
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: The analysis was performed on the Adapted persistence cohort, subset for MMR testing (Adapted ATP cohort for each specific time point).
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 410 | 409 | 137
mIU/mL
  Anti-measles, Year 4 | 3290.9 [3025.8 to 3579.2] | 1803.5 [1635.8 to 1988.5] | 1724.4 [1431.7 to 2077.0]
  Anti-measles, Year 6: number analyzed (Participants) | 406 | 221 | 137
  Anti-measles, Year 6 | 2795.9 [2544.7 to 3072.0] | 1727.7 [1514.3 to 1971.1] | 1369.0 [1125.7 to 1665.0]
  Anti-measles, Year 8: number analyzed (Participants) | 357 | 125 | 119
  Anti-measles, Year 8 | 2342.0 [2115.3 to 2593.0] | 1575.1 [1296.9 to 1913.1] | 1175.5 [963.6 to 1434.0]
  Anti-measles, Year 10: number analyzed (Participants) | 344 | 39 | 116
  Anti-measles, Year 10 | 1857.2 [1664.0 to 2072.8] | 997.5 [726.7 to 1369.1] | 913.6 [747.0 to 1117.4]

30. Secondary Outcome: Phase B: Number of Subjects With Anti-measles Antibody Concentrations Above the Cut-off Value
Description: The anti-measles antibody concentration cut-off value assessed was ≥ 150 mIU/mL, in the sera of subjects seronegative before vaccination.
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 410 | 409 | 137
Participants
  Anti-measles, Year 4 | 407 | 402 | 131
  Anti-measles, Year 6: number analyzed (Participants) | 406 | 221 | 137
  Anti-measles, Year 6 | 402 | 218 | 128
  Anti-measles, Year 8: number analyzed (Participants) | 357 | 125 | 119
  Anti-measles, Year 8 | 353 | 121 | 113
  Anti-measles, Year 10: number analyzed (Participants) | 344 | 39 | 116
  Anti-measles, Year 10 | 339 | 39 | 109

31. Secondary Outcome: Phase B: Immune Response to Mumps With Respect to Anti-mumps Antibody Concentrations
Description: as for outcome 8
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 407 | 407 | 136
U/mL
  Anti-mumps, Year 4 | 1088.9 [974.9 to 1216.3] | 905.3 [810.0 to 1011.9] | 1059.1 [878.9 to 1276.3]
  Anti-mumps, Year 6: number analyzed (Participants) | 398 | 217 | 132
  Anti-mumps, Year 6 | 999.7 [897.4 to 1113.7] | 920.5 [800.3 to 1058.8] | 1030.3 [879.1 to 1207.6]
  Anti-mumps, Year 8: number analyzed (Participants) | 348 | 120 | 117
  Anti-mumps, Year 8 | 875.7 [781.9 to 980.9] | 865.7 [718.3 to 1043.3] | 869.1 [723.3 to 1044.2]
  Anti-mumps, Year 10: number analyzed (Participants) | 339 | 37 | 115
  Anti-mumps, Year 10 | 889.3 [794.4 to 995.6] | 1054.0 [797.2 to 1393.6] | 912.7 [759.5 to 1096.8]

32. Secondary Outcome: Phase B: Number of Subjects With Anti-mumps Antibody Concentrations Above the Cut-off Value
Description: The anti-mumps antibody concentration cut-off value assessed was ≥ 231 U/mL, in the sera of subjects seronegative before vaccination.
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 407 | 407 | 136
Participants
  Anti-mumps, Year 4 | 368 | 357 | 123
  Anti-mumps, Year 6: number analyzed (Participants) | 398 | 217 | 132
  Anti-mumps, Year 6 | 360 | 196 | 127
  Anti-mumps, Year 8: number analyzed (Participants) | 348 | 120 | 117
  Anti-mumps, Year 8 | 305 | 107 | 108
  Anti-mumps, Year 10: number analyzed (Participants) | 339 | 37 | 115
  Anti-mumps, Year 10 | 305 | 36 | 108

33. Secondary Outcome: Phase B: Immune Response to Rubella With Respect to Anti-rubella Antibody Concentrations
Description: as for outcome 10
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 407 | 410 | 137
IU/mL
  Anti-rubella, Year 4 | 44.4 [40.9 to 48.3] | 50.8 [46.8 to 55.2] | 49.0 [42.9 to 55.9]
  Anti-rubella, Year 6: number analyzed (Participants) | 403 | 224 | 137
  Anti-rubella, Year 6 | 30.1 [27.9 to 32.4] | 34.0 [30.6 to 37.7] | 33.3 [29.2 to 37.9]
  Anti-rubella, Year 8: number analyzed (Participants) | 354 | 124 | 119
  Anti-rubella, Year 8 | 20.8 [19.0 to 22.9] | 26.7 [22.7 to 31.5] | 23.3 [19.8 to 27.3]
  Anti-rubella, Year 10: number analyzed (Participants) | 342 | 39 | 116
  Anti-rubella, Year 10 | 18.8 [17.0 to 20.7] | 29.2 [22.7 to 37.7] | 20.8 [17.6 to 24.6]

34. Secondary Outcome: Phase B: Number of Subjects With Anti-rubella Antibody Concentrations Above the Cut-off Value
Description: The anti-rubella antibody concentration cut-off value assessed was ≥ 4 IU/mL, in the sera of subjects seronegative before vaccination.
Time Frame: At Year 4, Year 6, Year 8 and Year 10 time points
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 407 | 410 | 137
Participants
  Anti-rubella, Year 4 | 407 | 408 | 137
  Anti-rubella, Year 6: number analyzed (Participants) | 403 | 224 | 137
  Anti-rubella, Year 6 | 402 | 222 | 136
  Anti-rubella, Year 8: number analyzed (Participants) | 354 | 124 | 119
  Anti-rubella, Year 8 | 347 | 120 | 116
  Anti-rubella, Year 10: number analyzed (Participants) | 342 | 39 | 116
  Anti-rubella, Year 10 | 334 | 39 | 112

35. Secondary Outcome: Phase B: Characteristics of Zoster Cases
Description: Zoster cases were characterized by number and character of lesions, duration of rash, incidence of fever, systemic signs, the assessment by investigator, complications, treatment, outcome and intensity of severity.
Time Frame: From 6 weeks after Dose 2 until study end (Year 10)
Population: The analysis was performed on the ATP Cohort for Efficacy (Phase A), which included all evaluable subjects who had efficacy follow-up starting from 42 days post dose 2 and from the period when Phase A was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | OKAH Group | MMR Group
Number analyzed (Participants) | 4 | 2
Participants
  Rash: number of lesions, 1-50 | 4 | 2
  Rash: number of lesions, 51-100 | 0 | 0
  Rash: number of lesions, 101-500 | 0 | 0
  Rash: number of lesions, 501+ | 0 | 0
  Character of most lesions, Macular | 0 | 0
  Character of most lesions, Papular | 2 | 1
  Character of most lesions, Vesicular | 2 | 1
  Character of most lesions, Haemorrhagic | 0 | 0
  Duration of rash, 0 days | 0 | 0
  Duration of rash, 1-5 days | 0 | 1
  Duration of rash, 6-10 days | 1 | 0
  Duration of rash, 11-15 days | 3 | 1
  Duration of rash, 16+ days | 0 | 0
  Max. number of lesions [investigator], 1-50 | 4 | 2
  Max. number of lesions [investigator], 51-100 | 0 | 0
  Max. number of lesions [investigator], 101-500 | 0 | 0
  Max. number of lesions [investigator], 501+ | 0 | 0
  Fever, No fever | 4 | 2
  Fever, 38.8°C to 39.9°C | 0 | 0
  Fever, 40+ °C | 0 | 0
  Systemic signs, Pain in back or abdomen | 2 | 1
  Systemic signs, Interstitial pneumonia | 0 | 0
  Systemic signs, Encephalitis | 0 | 0
  Assessment by investigator, Does not appear ill | 3 | 2
  Assessment by investigator, Moderately ill | 1 | 0
  Assessment by investigator, Severely ill | 0 | 0
  Complications, Yes | 0 | 0
  Complications, No | 4 | 2
  Treatment, Yes | 2 | 1
  Treatment, No | 2 | 1
  Outcome, Recovered/resolved | 4 | 2
  Outcome, Recovered/resolved with sequelae | 0 | 0
  Intensity of severity, Mild | 4 | 2
  Intensity of severity, Moderately severe | 0 | 0
  Intensity of severity, Severe | 0 | 0

36. Secondary Outcome: Phase B: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 21
Time Frame: From the beginning of Phase B (Year 2) up to study end (Year 10)
Population: The analysis was performed on the Total enrolled cohort in Phase B, which included all subjects from the Total Vaccinated cohort in Phase A who returned for at least one visit in Phase B
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 1961 | 1978 | 641
Participants | 290 | 317 | 93

37. Secondary Outcome: Phase B: Health Economics Analysis of Factors Leading to Indirect Costs Due to Varicella Illness
Description: as for outcome 22
Time Frame: During Phase B
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MMRV Group | OKAH Group | MMR Group
Number analyzed (Participants) | 38 | 227 | 150
Hours
  Time lost from work [hours] | 42.8 (44.1) | 44.6 (31.1) | 57.8 (36.8)
  Time lost for subjects [hours] | 40.7 (35.6) | 48.0 (34.1) | 57.2 (36.1)
  Time of requested assistance [hours] | 0 (0) | 45.7 (21.5) | 49.4 (50.0)

ADVERSE EVENTS:
Time Frame: Solicited local AEs: 4-days (Days 0-3) post dose 1 (Day 0) and dose 2 (Day 42). Solicited general and unsolicited AEs: 43-days (Days 0-42) post dose 1 (Day 0) and dose 2 (Day 42). Serious adverse events: From Day 0 up to the end of study (Year 10).
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed
Arm/Group | MMRV Group | OKAH Group | MMR Group
All-Cause Mortality (participants affected / at risk) | 1/2489 | 1/2487 | 0/827
Serious Adverse Events (participants affected / at risk) | 649/2489 | 681/2487 | 208/827
Other Adverse Events (participants affected / at risk) | 666/2489 | 641/2487 | 204/827
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMRV Group (N=2489) | OKAH Group (N=2487) | MMR Group (N=827)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 2 (2) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 7 (8) | 9 (9) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Long qt syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anomaly of external ear congenital (Congenital, familial and genetic disorders) | 1 (2) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Choledochal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Congenital oral malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 3 (3) | 3 (3) | 0 (0)
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Double ureter (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Duane's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hereditary pancreatitis (Congenital, familial and genetic disorders) | 0 (0) | 1 (5) | 0 (0)
Hernia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 8 (9) | 5 (5) | 0 (0)
Neurofibromatosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 12 (12) | 5 (5) | 2 (2)
Primary ciliary dyskinesia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Thalassaemia beta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Ear deformity acquired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
External ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Endocrine disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammation of lacrimal passage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 2 (2) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 14 (14) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 6 (6) | 0 (0)
Enteritis (Gastrointestinal disorders) | 6 (6) | 7 (7) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 31 (34) | 22 (25) | 9 (9)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 13 (13) | 16 (16) | 5 (6)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 6 (6) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1)
Accidental death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Crying (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia malignant (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Polyp (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (2) | 1 (1)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic oedema (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Atopy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2) | 1 (1)
Immunodeficiency (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
Adenoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 14 (14) | 12 (12) | 5 (5)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 47 (55) | 51 (65) | 15 (15)
Bronchitis haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 3 (3) | 9 (9) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Croup infectious (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Eczema impetiginous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 5 (5) | 5 (5) | 6 (6)
Enterobiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epstein-barr virus infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Erythema infectiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 67 (74) | 71 (79) | 26 (28)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 27 (27) | 42 (42) | 13 (13)
Gastroenteritis salmonella (Infections and infestations) | 2 (2) | 9 (9) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
H1n1 influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 5 (5) | 7 (7) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Laryngitis (Infections and infestations) | 39 (51) | 45 (56) | 8 (8)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Meningitis borrelia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Nasal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (17) | 6 (6) | 3 (3)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 3 (4) | 2 (2)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngitis fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 17 (19) | 7 (7) | 3 (3)
Otitis media acute (Infections and infestations) | 5 (5) | 7 (7) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Overgrowth bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Parvovirus b19 infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 4 (5) | 0 (0)
Pharyngitis (Infections and infestations) | 20 (21) | 13 (13) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 6 (6) | 10 (10) | 3 (3)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 70 (80) | 63 (66) | 30 (31)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pseudocroup (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (4) | 4 (4) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 7 (7) | 1 (1)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 3 (4) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 6 (6) | 2 (2) | 1 (1)
Scarlet fever (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 7 (7) | 4 (5) | 5 (5)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 23 (23) | 18 (19) | 7 (9)
Tonsillitis bacterial (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Toxocariasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 9 (9) | 4 (5) | 3 (4)
Tracheobronchitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Tuberculosis of intrathoracic lymph nodes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 9 (9) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (3) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 4 (4) | 11 (11) | 4 (4)
Viral myositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 5 (6) | 9 (10) | 5 (5)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 4 (4) | 10 (10) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Burn oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Chemical injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Child maltreatment syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 23 (24) | 26 (26) | 7 (8)
Contusion (Injury, poisoning and procedural complications) | 15 (15) | 13 (13) | 2 (2)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 6 (6) | 9 (9) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 3 (3) | 2 (3) | 2 (2)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 8 (8) | 9 (9) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 5 (5) | 9 (9) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Kidney contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Liver contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Pancreatic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Penile contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Struck by lightning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 6 (6) | 9 (9) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Venomous sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Medical observation (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 9 (10) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (6) | 3 (3) | 1 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 1 (4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 2 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rickets (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Autism (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Benign rolandic epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgraphia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyslexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 4 (5) | 5 (6) | 1 (2)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 21 (23) | 20 (23) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1)
Intellectual disability (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Language disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 5 (6) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 3 (3) | 3 (5) | 0 (0)
Breath holding (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Enuresis (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Learning disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Neurosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Reading disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Glomerulonephritis acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 3 (3) | 4 (4) | 1 (1)
Penis disorder (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0)
Testicular appendage torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular retraction (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 111 (116) | 123 (129) | 39 (39)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 8 (8) | 5 (5)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 3 (3)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Circumcision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.98% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMRV Group (N=2489) | OKAH Group (N=2487) | MMR Group (N=827)
Injection site erythema (General disorders) | 244 (325) | 183 (260) | 43 (60)
Pyrexia (General disorders) | 604 (849) | 574 (790) | 188 (253)
Injection site pain (General disorders) | 124 (165) | 111 (146) | 31 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.